CLINICAL TRIAL: NCT06125431
Title: Factors That Affect Trust Between Physicians and Patients
Status: Recruiting | Type: Observational
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Other Study IDs: 5230221
Record Dates: First submitted 2023-11-04; First posted 2023-11-09 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Trust

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this study is to evaluate patient perception and preference in physician attire. Eligible subjects admitted to medical-surgical hospital unit will complete a survey expressing perceptions and preference regarding physician attire.

DETAILED DESCRIPTION:
Hospitalists (internal medicine physicians) work in one week rotations. Each hospitalist will serve as a control.

During one week rotation, the hospitalist will wear surgical scrubs throughout the rotation. At the end of the rotation (or prior to subject discharge, whichever occurs first), the hospitalist will ask subjects seen during that rotation to complete the survey regarding the hospitalist attire.

During a second week of rotation, the hospitalist will wear professional attire with a white coat throughout that rotation. At the end of the rotation (or prior to subject discharge, whichever occurs first), the hospitalist will ask subjects seen during that rotation to complete the survey regarding the hospitalist attire.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18 years of ages or older
* Admitted to LLUMC medical surgical unit, under care of internal medicine physician
* Primary language is English or Spanish

Exclusion Criteria:

* Less than 18 years of age
* altered mental status or severe dementia
* Hearing or vision impairment that would preclude subject from completing survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized internal medicine patients, 18 years and older, with English or Spanish as primary language.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Patient Preference for Type of Physician Attire | At the end of hospitalist rotation or prior to subject discharge, whichever occurs first, not to exceed one week from study enrollment.
  Subjects will complete a one-time survey via paper or iPAD. The survey is based on the Modified Trust in Physician Scale: A Measure to Assess Interpersonal Trust in Patient Physician Relationships with answers provided on a 5 point Likert Scale where 1 means strongly disagree, 2 means disagree, 3 is neutral, 4 means agree and 5 means strongly agree. The total score will reflect patient preference for traditional physician attire (street clothes and white coat) or casual physician attire (surgical scrubs). A high score would reflect a favorable response for the physician wearing traditional attire.

CONTACTS AND LOCATIONS:
Locations (1):
- Loma Linda University Medical Center, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No